CLINICAL TRIAL: NCT06018155
Title: Study of the Relation Between the Fat Infiltration of the Multifidus Muscle and the Lumbar Foraminal Stenosis, by 2D and 3D Segmentation
Acronym: FIMFos
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Neuro02
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Degenerative Condition, Neurologic
MeSH Terms: conditions — Low Back Pain; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single cohort: Cohort of patients suffering from low back pain and candidate to a spine surgery included in a database previously constituted
  Interventions: Other: Spine surgery

INTERVENTIONS:
Other: Spine surgery — Cohort of patients suffering from low back pain and candidate to a spine surgery included in a database previously constituted

SUMMARY:
The aim of this study is to evaluate the correlation between the fat infiltration of the lumbar multifidus muscle and several parameters including the severity of the lumbar foraminal stenosis. The investigators will analyse lumbar MRI of patients previously included in a database of patients suffering from low back pain. Foraminal stenosis, muscle fat infiltration and other imaging lumbar parameters will be studied by 2D and 3D manuel segmentation, semi-automatic segmentation. Correlations between factors influencing the muscle fat infiltration will be studied by univariate and multivariate statistical analysis.

ELIGIBILITY:
Patients suffering from low back pain and candidate to a spine surgery included in a database previously constituted, for who the following parameters are available: lumbar 3D MRI with T2 weighted sequences, informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from low back pain and candidate to a spine surgery included in a database previously constituted
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of muscle fat infiltration | 1 year
  Muscle fat infiltration (%) will be evaluated by 2D segmentation analysis of T2 weighted lumbar spine MRIs
Percentage of muscle fat infiltration | 1 year
  Muscle fat infiltration (%) will be evaluated by 3D segmentation analysis of T2 weighted lumbar spine MRIs

SECONDARY OUTCOMES:
Lumbar foraminal stenosis | 1 year
  Lumbar foraminal stenosis will be evaluated by 2D segmentation analysis of T2 weighted lumbar spine MRIs and expressed as a nerve/foramen surface ratio, and by the Lee et al. Classification

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No